CLINICAL TRIAL: NCT07205757
Title: Adding Lidocaine to Custodiol® Cardioplegia to Decrease Post-bypass Ventricular Arrhythmias in Adult Patients Undergoing Coronary Artery Bypass Grafting (CABG) Surgery; A Prospective Randomized Double-Blinded Clinical Trial.
Brief Title: Adding Lidocaine to Custodiol Mixture
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Hasan Ragab, Lecturer of Anesthesiology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R 751
Record Dates: First submitted 2025-09-18; First posted 2025-10-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: CAD; Arrhythmia Ventricular
Keywords: Custodiol; lidocaine; Bretschneider solution; Ventricular arrythmia
MeSH Terms: interventions — Lidocaine; Bretschneider cardioplegic solution

STUDY DESIGN:
Intervention Model Description: This randomized double-blinded clinical trial will be reported following the tenets of the Declaration of Helsinki and the Consolidated Standards of Reporting Trials (CONSORT) 2025-updated statement.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized into two equal groups (1:1 allocation) using a computer-generated random number that will be enclosed in a sealed opaque envelope opened by an anesthesiologist, who is responsible for preparing the cardioplegia solution outside the OR and will not be involved in patient management or data collection.
  Patients, cardiothoracic surgeons, anesthesiologists, and data collectors will be blinded to group allocation until the end of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custodiol group (Active Comparator): standard Custodiol cardioplegia solution (manufactured by Dr. Franz Köhler Chemie GmbH, Bensheim, Germany), punctured at the injection port with a 10-cc syringe for blinding
  Interventions: Drug: Custodiol Solution
- Lidocaine and Custodiol group (Experimental): the modified solution prepared by adding 6.5 ml of 2% lidocaine (Lidocaine HCL -Sunny Pharmaceutical) to each 1 L bag of Custodiol (Group L), using a 10-cc syringe.
  Interventions: Drug: Lidocaine Hydrochloride; Drug: Custodiol Solution

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — 6.5 ml of 2% lidocaine (Lidocaine HCL -Sunny Pharmaceutical)
  Other Names: Xylocaine
  Arms: Lidocaine and Custodiol group
Drug: Custodiol Solution — cardioplegia solution will be administered as a single dose of 20 mL/kg over 6-8 minutes at a temperature of 5-8 °C. An additional half dose of the same solution will be prepared and infused if the procedure exceeds 180 minutes after the initial dose is completed.
  Other Names: Bretschneider solution; HTK solution

SUMMARY:
The Bretschneider solution, also known as Custodiol, has been widely used in open-heart surgery requiring cardiopulmonary bypass (CPB) since its introduction in 1970. Custodiol is widely favored by cardiac surgeons, being administered as a single dose, and is supposed to offer myocardial protection for up to three hours, permitting an uninterrupted surgical time, especially for intricate procedures The literature continues to debate the superiority of custodial and other cardioplegic solutions, such as the Del Nido and St. Thomas solutions, regarding both short-term and long-term outcomes. Clinical trials and daily practice showed that the use of custodial cardioplegic solution is associated with increased incidences of ventricular arrhythmias, and subsequently, the use of a defibrillator after Aortic Cross Clamp (ACC) removal at the end of CPB when compared to other types of cardioplegia solutions .One of the reasons for this difference mentioned in the literature is the lidocaine contained in other types of cardioplegic solutions. Lidocaine acts as a membrane stabilizer by blocking rapid sodium channels in the heart, thus preventing arrhythmias, in addition to its ability to inhibit calcium influx, which is the primary cause of ischemic-reperfusion injury.

Based on these data, the investigators hypothesize that the increased incidence of Ventricular arrhythmias with the use of Custodiol compared to other solutions, such as St Thomas and Del Nido, may be attributed to the absence of lidocaine. Although Custodiol contains tryptophan as a membrane-stabilizing component, it may be beneficial to add lidocaine to the Custodiol mixture to decrease the incidence of VF after cross-clamp removal in adult patients undergoing elective CABG.

DETAILED DESCRIPTION:
After Ethical Review Board of Fayoum University Hospital (FUH) approval and clinicaltrials.gov registration, all patients scheduled for isolated on-pump Coronary Artery Bypass Grafting (CABG) surgery in FUH starting from August 2025 will be enrolled in the study by signing a written informed consent until the sample size is fulfilled. This randomized double-blinded clinical trial will be reported following the tenets of the Declaration of Helsinki and the Consolidated Standards of Reporting Trials (CONSORT) 2025-updated statement.

Patients will be randomized into two equal groups (1:1 allocation) using a computer-generated random number that will be enclosed in a sealed opaque envelope opened by an anesthesiologist, who is responsible for preparing the cardioplegia solution outside the OR and will not be involved in patient management or data collection.

According to each envelope, the Study solution will be either standard Custodiol cardioplegia solution (manufactured by Dr. Franz Köhler Chemie GmbH, Bensheim, Germany), punctured at the injection port with a 10-cc syringe for blinding (Group C), or the modified solution prepared by adding 6.5 ml of 2% lidocaine (Lidocaine HCL -Sunny Pharmaceutical) to each 1 L bag of Custodiol (Group L), using a 10-cc syringe. According to the patient's weight, one or two 1-L solutions will be prepared (calculated at 20 ml/kg, with a maximum of 2 L), kept at 5-8°C, and handed to the cardiothoracic anesthesia team when ordered. Patients, cardiothoracic surgeons, anesthesiologists, and data collectors will be blinded to group allocation until the end of the study.

All patients will be preoperatively examined and investigated by complete blood count, coagulation profile, liver and kidney functions, and electrolytes. A chest x-ray, Electrocardiography (ECG), echocardiography, Carotid arterial duplex, and Coronary angiography will be routinely ordered. Patients will receive an intramuscular injection of 10 mg morphine on the morning of the operation Upon arrival at OR, Standard monitoring will be applied, involving a 5-lead ECG and pulse oximetry. Blood pressure will be monitored through a 20-G cannula inserted into either the right or left radial artery under local anesthesia. Atracurium (0.5 mg/kg), midazolam (2-5 mg), fentanyl (2-5 μg/kg), and propofol (1-2 mg/kg) will be used to induce general anesthesia following pre-oxygenation.

After tracheal intubation, patients will be mechanically ventilated with an Oxygen and air mixture, maintaining normocapnia confirmed by capnogram and arterial blood gas analysis. A urinary catheter, an esophageal temperature probe, and a right internal jugular triple-lumen central venous catheter will be inserted. Inhalational isoflurane (0.4 to 1 %) and atracurium infusion at 0.5 mg/kg/h will be used to maintain anesthesia and muscle relaxation. A 50-100 µg/kg/min propofol infusion will replace isoflurane inhalation during extracorporeal circulation.

To achieve an active clotting time of greater than 480 seconds, patients will receive intravenous heparin (300-500 units/kg body weight) prior to the initiation of cardiopulmonary bypass (CPB). An ascending aortic cannula and a two-stage right atrial cannula will be used to implement CPB. Before, during, and following CPB, mean arterial pressure will be adjusted to be higher than 60 mmHg (pump blood flow: 2.4 l/min/m2).

Myocardial protection:

The antegrade approach will be utilized to deliver the cardioplegic solution through the coronary ostia or the aortic root, as appropriate. The cardioplegic solution will be either the classic Custodiol or the modified Custodiol according to the group allocation of each patient.

A ready-blinded cardioplegia solution will be administered as a single dose of 20 mL/kg over 6-8 minutes at a temperature of 5-8 °C. An additional half dose of the same solution will be prepared and infused if the procedure exceeds 180 minutes after the initial dose is completed.

Mean arterial blood pressure will be maintained at 50-70 mmhg during the bypass period.

By completing distal anastomosis and before the ACC removal, all patients will be rewarmed to a core temperature of 36°C and have an arterial blood gas analysis that should have a normal PH (7.35-7.45), a normal potassium level (3.5 - 5.5) mg/dl, and a hemoglobin level above 10 g/dl, any abnormal value should be corrected before ACC removal. A 1.5 mg/kg lidocaine and 1 gram of Magnesium sulfate will be administered on the cardiopulmonary bypass machine just before the ACC release.

After cross clamp removal, internal paddles will be used to defibrillate any ventricular fibrillation VF with 10 joule of energy.

If VF is resistant after three 10 j shocks, a 150 mg of Amiodarone will be administered and subsequent defibrillator shocks with escalating energy level 10, 20, and 30 joules will be used.

Proximal venous graft anastomoses will be carried out after applying a partial aortic cross clamp. Then, the patient will be gradually weaned from cardiopulmonary bypass after rewarming to normal core temperature and applying any needed inotropic or vasopressor support to maintain optimal cardiac output.

Protamine sulfate will be administered after achieving hemodynamic stability to reverse the actions of heparin. The patient will be transferred to the postoperative cardiac surgery intensive care unit after completing hemostasis, drains, epicardial pacing wires, and wound closure.

Sample size calculation:

the sample size was calculated based on a previous study from Kammerer et.al, the incidence of ventricular fibrillation after ACC removal with Custodiol was 45.45 % and the incidence with conventional cardioplegic solution was 9.6 %. the investigators hypothesize that the addition of lidocaine to Custodiol will decrease the incidence of VF after ACC removal to a percentage similar to the conventional cardioplegic solution.

To account for this proportion difference, a minimal sample size of 31 patients in each group is needed to get a power level of 0.90 and an alpha level of 0.05. The calculated sample size will be increased to 35 in each group to allow for dropouts up to 10%. IBM SPSS software version 31 was used to estimate the required sample size.

Statistical Analysis Statistical analysis will be performed using IBM SPSS software version 31. Descriptive statistics will be used to summarize participant demographics and clinical characteristics. Continuous variables will be reported as means ± standard deviations or medians with interquartile ranges, depending on normality of data assessed using the Shapiro-Wilk test. Categorical variables will be presented as frequencies and percentages. Independent t-tests or Mann-Whitney U tests will be applied to compare continuous variables between the two groups, while chi-square or Fisher's exact tests will be used for categorical variables as appropriate. Survival analysis with Kaplan Meier plot will be used for comparison of time to event variables. P-value less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective Coronary artery bypass grafting surgery

Exclusion Criteria:

* Emergency or Redo surgery.
* Baseline rhythm other than sinus rhythm
* Any degree of heart block, bundle branch block or hemiblock
* Known allergy to lidocaine.
* Chronic kidney disease.
* Hepatic impairment.
* Severe psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
incidence of ventricular fibrillation (VF) | Perioperative
  incidence of VF occurring after Aorta cross-clamp (ACC) removal

SECONDARY OUTCOMES:
Troponin I (µg/L) | At immediate postoperatively, 12 and 24 hours postoperative
  Troponin I to assess myocardial protection between the two cardioplegia solutions used.
Number of defibrillator shocks | Perioperative
  shocks required to terminate ventricular arrhythmia after ACC removal
Total volume of cardioplegia solution (in ml). | Perioperative
  cardioplegia volume given to the patient
Total cross-clamp time | from cross clamp until removal of aorta cross clamp up to 6 hours
  in minutes
total CPB time | from starting CPB until weaning from bypass is completed up to 6 hours
  in minutes
Number of grafts | at the end of surgery up to 6 hours
  anastomosis coronary grafts
Time taken to cardiac arrest after cardioplegia infusion | from the start of cardioplegia administration until asystole up to one hour
  time to asystole
Left ventricular ejection fraction assessed both preoperative and after 24 hours postoperatively. | assessed both preoperative and after 24 hours postoperatively.
  echo assessment
Preoperative EURO II score | assessed preoperatively at the start of patient enrollment
  EURO II score
Inotropic support. | assessed after patient is transferred to intensive care up to 6 hours from start of surgery
  the need for inotropes on transfer to intensive care
Total time of inotropes or vasopressor requirement in hours | assessed after patient is weaned from inotropes up to one month
  the need for inotropes in intensive care
CK-MB (U/L) . | at immediate postoperatively, 12 and 24 hours after surgery
  CK-MB (U/L) .
Serum lactate level | at immediate postoperatively, 12 and 24 hours after surgery.
  Serum lactate level
Incidence of postoperative Myocardial infarction | assessed from icu admission until discharge up to one month
  Incidence of postoperative Myocardial infarction
Incidence of postoperative Atrial fibrillations | assessed from icu admission until ICU discharge up to one month
  Incidence of postoperative Atrial fibrillations
Time for weaning from mechanical ventilation | assessed from icu admission until ventilator weaning up to one month
  from mechanical ventilation (in hours).
ICU length of stay | assessed from icu admission until ICU discharge up to one month
  in hours
hospital length of stay (in days) | assessed from icu admission until home discharge up to one month
  in days
Mortality rate | assessed up to one month postoperatively
  Mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Ragab, MD, Principal Investigator — Lecturer of Anesthesiology
Locations (1):
- Fayoum University Hospital, Al Fayyum, Egypt

REFERENCES:
- [Background] Bretschneider HJ, Hubner G, Knoll D, Lohr B, Nordbeck H, Spieckermann PG. Myocardial resistance and tolerance to ischemia: physiological and biochemical basis. J Cardiovasc Surg (Torino). 1975 May-Jun;16(3):241-60. PMID 239002
- [Background] Barbero C, Pocar M, Marchetto G, Cura Stura E, Calia C, Dalbesio B, Filippini C, Salizzoni S, Boffini M, Rinaldi M, Ricci D. Single-Dose St. Thomas Versus Custodiol(R) Cardioplegia for Right Mini-thoracotomy Mitral Valve Surgery. J Cardiovasc Transl Res. 2023 Feb;16(1):192-198. doi: 10.1007/s12265-022-10296-z. Epub 2022 Aug 8. PMID 35939196
- [Background] Ferguson ZG, Yarborough DE, Jarvis BL, Sistino JJ. Evidence-based medicine and myocardial protection--where is the evidence? Perfusion. 2015 Jul;30(5):415-22. doi: 10.1177/0267659114551856. Epub 2014 Oct 8. PMID 25298053
- [Background] Chan J, Oo S, Butt S, Benedetto U, Caputo M, Angelini GD, Vohra HA. Network meta-analysis comparing blood cardioplegia, Del Nido cardioplegia and custodiol cardioplegia in minimally invasive cardiac surgery. Perfusion. 2023 Apr;38(3):464-472. doi: 10.1177/02676591221075522. Epub 2022 Feb 27. PMID 35225070
- [Background] Ghiragosian C, Harpa M, Stoica A, Sanziana FO, Balau R, Hussein HA, Elena GS, Neagoe RM, Suciu H. Theoretical and Practical Aspects in the Use of Bretschneider Cardioplegia. J Cardiovasc Dev Dis. 2022 Jun 2;9(6):178. doi: 10.3390/jcdd9060178. PMID 35735807
- [Background] Kantathut N, Luangpatom-Aram K, Khajarern S, Leelayana P, Cherntanomwong P. Comparison of Single-Dose Cardioplegia in Valvular Heart Surgery: Lactated Ringer's-Based del Nido vs. Histidine-Tryptophan-Ketoglutarate Cardioplegia Solution. Braz J Cardiovasc Surg. 2023 Oct 6;38(6):e20220447. doi: 10.21470/1678-9741-2022-0447. PMID 37801520
- [Background] Duan L, Hu GH, Wang E, Zhang CL, Huang LJ, Duan YY. Del Nido versus HTK cardioplegia for myocardial protection during adult complex valve surgery: a retrospective study. BMC Cardiovasc Disord. 2021 Dec 18;21(1):604. doi: 10.1186/s12872-021-02411-w. PMID 34922443
- [Background] Hearse DJ, O'Brien K, Braimbridge MV. Protection of the myocardium during ischemic arrest. Dose-response curves for procaine and lignocaine in cardioplegic solutions. J Thorac Cardiovasc Surg. 1981 Jun;81(6):873-9. PMID 7230856
- [Background] Siddiqi S, Blackstone EH, Bakaeen FG. Bretschneider and del Nido solutions: Are they safe for coronary artery bypass grafting? If so, how should we use them? J Card Surg. 2018 May;33(5):229-234. doi: 10.1111/jocs.13539. Epub 2018 Feb 14. PMID 29444545